CLINICAL TRIAL: NCT06449937
Title: Analysis of the Efficacy of Local Liver Treatment for Multi-organ Colorectal Cancer Metastases: A Prospective, Multicenter, Non-randomized Concurrent Controlled Study
Brief Title: Local Liver Treatment for Multi-organ Colorectal Cancer Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024KY109
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Colorectal Carcinoma; Multi-organ Metastatic Colorectal Cancer; Metastatic Malignant Neoplasm in the Liver
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Radical local treatment combined with systematic treatment) (Experimental): Patients undergo radical local treatment of liver metastases (hepatectomy, ablation) combined with systematic treatment.
  Interventions: Procedure: Radical local Surgery; Drug: Systemic therapy
- Group II (systematic treatment only or combined with local interventional therapy) (Active Comparator): Patients undergo systemic therapy only or combined with local interventional therapy (TACE, HAIC).
  Interventions: Drug: Systemic therapy; Other: Interventional therapy

INTERVENTIONS:
Procedure: Radical local Surgery — Radical local resection of liver metastases ( hepatectomy, ablation )
  Arms: Group I (Radical local treatment combined with systematic treatment)
Drug: Systemic therapy — Chemotherapy, targeted drug therapy, immunotherapy treatment.
  Other Names: Chemotherapy, Cancer, General; Targeted therapy; immunotherapy
Other: Interventional therapy — Transcatheter arterial chemoembolization (TACE) Hepatic arterial infusion chemotherapy (HAIC)
  Arms: Group II (systematic treatment only or combined with local interventional therapy)

SUMMARY:
The purpose of this study was to investigate the effect of only local radical treatment of liver metastases combined with systematic treatment in the treatment of patients with multiple organ metastases of colorectal cancer, whether it can benefit the prognosis and explore the risk factors related to the prognosis.

DETAILED DESCRIPTION:
Primary objective:

1.To determine the survival benefit of local radical resection of liver metastases in patients with resectable liver and controllable extrahepatic metastases from colorectal cancer.

Secondary objectives:

1. To explore the prognosis-related risk factors in patients with colorectal cancer liver metastases combined with extrahepatic metastases
2. To assess patients' quality-of-life in each treatment group with questionnaires.
3. To evaluate the safety of the treatment in each treatment group.

Grouping Method: Patients are assigned to 1 of 2 groups according to their willingness.

GROUP I: Patients undergo radical local treatment of liver metastases (hepatectomy, ablation) combined with systemic therapy.

GROUP II: Patients receive Systemic therapy only or combined local interventions (TACE, HAIC)

Patients are followed up every 3 months up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-80 years of age.
* Patients volunteered to join the study and signed informed consent, with good compliance and follow-up.
* Primary colorectal tumors can be radically resected or resected and histopathologically diagnosed as colorectal cancer.
* Patients with synchronous or metachronous diagnosis of liver metastasis and extrahepatic metastasis by computed tomography (CT) or magnetic resonance imaging (MRI).Extrahepatic metastases are stable and controllable as determined by Multi-disciplinary Treatment (MDT).
* Patients receive only first- or second-line systemic therapy.
* Radical local treatment can be performed after MDT evaluation, and the indications at least meet the following one:

  * Hepatectomy: liver metastases can be completely (R0) removed and required to retain sufficient functional liver tissue;
  * Ablation therapy: The maximum diameter of liver metastases<3 cm, and the maximum number of ablation ≤ 5.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy of at least 3 months.
* Child-Pugh score ≤ 7.
* Laboratory routine examination (blood routine, liver and kidney function, coagulation function, etc.) no significant abnormalities:

  * Absolute neutrophil count (ANC) ≥ 1.5×10^9/l;
  * Platelet count (PLT) ≥ 100*10^9/l;
  * Hemoglobin ≥ 9g/dl;
  * TBIL<1.5 times the upper limit of normal (ULN);
  * ALT and AST< 5*ULN;
  * Serum creatinine ≤ 1.5 * ULN or Creatinine clearance> 50 ml/min;
  * Albumin > 30 g/l.

Exclusion Criteria:

* Patients with only liver metastasis confirmed by CT or MRI.
* History of hepatic encephalopathy or liver transplantation.
* Evidence of brain metastases.
* Pregnant or breast-feeding women.
* History of other malignant tumors (except thyroid cancer and carcinoma in situ) can be included in the study if the individual has remained disease-free for at least 5 years.
* Patients with acute cardiovascular and cerebrovascular diseases such as acute cerebral infarction and acute coronary syndrome within 1 month, and the cardiovascular clinical symptoms or diseases were not well controlled.
* NYHA class 3-4 or left ventricular ejection fraction (LVEF) < 50 % by echocardiography.
* Uncontrollable hypertension, blood pressure > 160 / 95 mmHg after treatment, history of hypertensive crisis or hypertensive encephalopathy.
* Uncontrollable infection > grade 2 (NCI-CTC version 5.0).
* Patients with respiratory insufficiency : PaO2 < 60 mmHg at rest , with or without PaCO2 > 50 mmHg.
* Patients with a large amount of ascites (ultrasound examination showed an echoless area around the liver and spleen, pelvic cavity, and intestinal loops, and the mesentery and intestinal canal were seen floating in the echoless area ) or malignant ascites (cancer cells were found in ascites or ascites CEA was higher than peripheral blood).
* Coagulation dysfunction ( INR > 1.5 or APTT > 1.5*ULN ), with bleeding tendency.
* Long-term unhealed wounds or fractures, major surgery or severe traumatic injury, fracture or ulcer occurred within 4 weeks.
* Patients with a history of mental drug abuse and who could not quit or had mental disorders.
* According to the investigator's judgment, patients with concomitant diseases that seriously endanger patient safety or affect patient completion of the study.
* According to the investigator's judgment, patients who are not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of study inclusion until the date of death or or the date of last follow-up, assessed up to 2 years
  Differences in overall survival between the two arms were assessed using the log-rank test; Cox proportional hazards regression models were used to determine the factors and hazard ratios associated with overall survival.

SECONDARY OUTCOMES:
Liver-specific progression free survival rates | Date of study inclusion to until local recurrence or progression in the liver or death from any cause, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate time to intrahepatic recurrence or progression or death from any cause in patients.
Incidence of adverse events | Assessed up to 2 years
  Record the frequency and percentage of adverse events, their grade, and their relationship to radical local treatment.
Quality of life scores-EORTC QLQ-C30 (version 3) questionnaire | Assessed up to 2 years
  Summarized using descriptive statistics, including mean, standard deviation, median and range.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Zhou Wang, MD PhD, Study Director — Anhui province hospital; Xiao-Ming Wang, MD PhD, Principal Investigator — First Affiliated Hospital of Wannan Medical College; Yu-Zhi Hu, MD, Principal Investigator — The Second People's Hospital of Wuhu; Yi-Ming Cao, MD, Principal Investigator — Ma'anshan People's Hospital; Qing-Song Yang, MD, Principal Investigator — The First People's Hospital of Chu Zhou; Si-Hua Wu, MD, Principal Investigator — Fuyang Cancer Hospital
Locations (6):
- China (6):
  - The First People's Hospital of Chu Zhou, Chuzhou, Anhui
  - Fuyang Cancer Hospital, Fuyang, Anhui
  - Anhui province hospital, Hefei, Anhui
  - Ma'anshan People's Hospital, Ma’anshan, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - The Second People's Hospital of Wuhu, Wuhu, Anhui

IPD SHARING:
Plan to Share IPD: No